CLINICAL TRIAL: NCT00082381
Title: Effect of AC2993 (Synthetic Exendin-4) Compared With Insulin Glargine in Patients With Type 2 Diabetes Also Using Combination Therapy With Sulfonylurea and Metformin
Brief Title: Effect of AC2993 Compared With Insulin Glargine in Patients With Type 2 Diabetes Also Using Combination Therapy With Sulfonylurea and Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H8O-MC-GWAA
Record Dates: First submitted 2004-05-06; First posted 2004-05-11 (Estimated); Results first posted 2013-07-31 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes; Insulin glargine; comparator; Amylin; Lilly
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Exenatide; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide Arm (Experimental): exenatide subcutaneous injection, twice daily; 5 mcg for 4 weeks followed by 10 mcg for 22 weeks
  Interventions: Drug: Exenatide (AC2993)
- Insulin Glargine Arm (Active Comparator): subcutaneous injection, once daily; forced titration to target blood glucose level
  Interventions: Drug: Insulin glargine

INTERVENTIONS:
Drug: Exenatide (AC2993) — subcutaneous injection, twice daily; 5 mcg for 4 weeks followed by 10 mcg for 22 weeks
  Other Names: Byetta
  Arms: Exenatide Arm
Drug: Insulin glargine — subcutaneous injection, once daily; forced titration to target blood glucose level
  Other Names: Lantus
  Arms: Insulin Glargine Arm

SUMMARY:
This is a multicenter, comparator-controlled, open-label, randomized, two-arm, parallel trial to compare the effect of exenatide twice daily and insulin glargine on glycemic control, as measured by hemoglobin A1c (HbA1c).

ELIGIBILITY:
Inclusion Criteria:

* Patients have been treated with a stable dose of one of the following for at least 3 months prior to screening: 1. 1500 to 2550 mg/day immediate-release metformin (or 1500 to 2000 mg/day extended-release metformin) and at least an optimally effective dose of a sulfonylurea, or 2. a fixed-dose sulfonylurea/metformin combination therapy with the same sulfonylurea and metformin requirements as for the individual components.
* HbA1c between 7.0% and 10.0%, inclusive.
* History of stable body weight (not varying by >10% for at least three months prior to screening).
* Female patients are not breastfeeding, and female patients of childbearing potential (not surgically sterilized and between menarche and 1-year postmenopause)

Exclusion Criteria:

* Patients are investigator site personnel directly affiliated with the study, or are immediate family of investigator site personnel directly affiliated with the study.
* Patients are employed by Lilly or Amylin.
* Patients have participated in this study previously or any other study using AC2993 or GLP-1 analogs.
* Patients have participated in an interventional medical, surgical, or pharmaceutical study within 30 days prior to screening. This criterion includes drugs that have not received regulatory approval for any indication at the time of study entry.
* Patients have had greater than three episodes of severe hypoglycemia within 6 months prior to screening.
* Patients are undergoing therapy for a malignancy, other than basal cell or squamous cell skin cancer.
* Patients have cardiac disease that is Class III or IV, according to the New York Heart Association criteria.
* Patients have a known allergy or hypersensitivity to insulin glargine, AC2993, or excipients contained in these agents.
* Patients have characteristics contraindicating metformin or sulfonylurea use, according to product-specific label, in the opinion of the investigator.
* Patients have a history of renal transplantation or are currently receiving renal dialysis or have serum creatinine >=1.5 mg/dL for males and >=1.3 mg/dL for females.
* Patients have obvious clinical signs or symptoms of liver disease, acute or chronic hepatitis, or alanine aminotransferase/serum glutamicpyruvic transaminase greater than three times the upper limit of the reference range.
* Patients have known hemoglobinopathy or chronic anemia.
* Patients are receiving chronic (lasting longer than 2 weeks) systemic glucocorticoid therapy (excluding topical and inhaled preparations) or have received such therapy within 2 weeks immediately prior to screening.
* Patients have used any prescription drug to promote weight loss within 3 months prior to screening.
* Patients have any other condition (including known drug or alcohol abuse or psychiatric disorder) that precludes them from following and completing the protocol, in the opinion of the investigator.
* Patients fail to satisfy the investigator of suitability to participate for any other reason.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2003-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, MD, Study Director — Eli Lilly and Company
Locations (91):
- United States (21):
  - Radiant Research-San Diego, San Diego, California
  - Dorothy L. and James E. Frank Diabetes Research Institute, San Mateo, California
  - Internal Medicine Associates Department of Research, Fort Myers, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Baptist Diabetes Associates, Miami, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Springfield Diabetes & Endocrine Center, Springfield, Illinois
  - Frederick Primary Care Associates, Frederick, Maryland
  - Radiant Research, Inc., St Louis, Missouri
  - Lovelace Scientific Resources, Inc., Las Vegas, Nevada
  - Diabetes, Endocrine & Nutrition, Hampton, New Hampshire
  - Lovelace Scientific Resources, Albuquerque, New Mexico
  - Great Lakes Medical Research, Westfield, New York
  - DOCS, Beth Israel Medical Center, Yonkers, New York
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Jon Shapiro, MD, Philadelphia, Pennsylvania
  - Endocrinology Consultants of East Tennessee, Knoxville, Tennessee
  - Israel Hartman, MD, Arlington, Texas
  - Diabetes & Glandular Research Associates, P.A., San Antonio, Texas
  - Jack Wahlen, MD, Ogden, Utah
  - Rainier Clinical Research Center, Inc., Renton, Washington
- Australia (10):
  - Australian Clinical Research Centre, Miranda, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Clinical Trial and Research Unit, Wollongong, New South Wales
  - Royal Brisbane Hospital, Brisbane, Queensland
  - Royal Adelaid Hospital, Adelaid, South Australia
  - Repatriation General Hospital, Daw Park, South Australia
  - SA Endocrine Clinical Research, Keswick, South Australia
  - Eastern Health (Box Hill Hospital), Box Hill, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Freemantle Hospital, Freemantle, Western Australia
- Belgium (6):
  - UZ Antwerpen, Endegem
  - UZ Gent, Ghent
  - UZ Gasthuisberg, Leuven
  - CHU Sart Tilman, Liège
  - A.Z. Jan Palfijn, Merksem
  - Sint Niklaasstraat, Sint-Gillis-Waas
- Brazil (4):
  - Hospital Nossa Senhora das Gracas, Curitiba
  - Centro Integrado de Diabetes e Hipertensao, Fortaleza
  - Centro de Pesquisas em Diabetes e Doencas Endocrino Metabolicas/HUWC/UFC, Fortaleza
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre
- Finland (3):
  - Eiran Sairaala c/o9 Clires, Helsinki
  - Torikeskuksen Laakariasema, Yliopistonkatu, Jyväskylä
  - Oulu Deakoness Institution, Oulu
- Germany (8):
  - Diabetologische Schwerpunktpraxis, Aschaffenburg
  - Diabetologische Scherpunktpraxis, Bosenheim
  - Diabetologische Schwerpunktpraxis, Dortmund
  - Krankenhaus Bethanien, Hamburg
  - Universitatskliniken des Saarlandes, Homburg/Saar
  - IKFE GmbH, Mainz
  - Profil Institut fur Stoffwechselforschung GmbH, Neuss
  - Diabetologische Schwerpunktpraxis, Neuwied
- Netherlands (5):
  - Diabetes Centrum Bilthoven, Bilthoven
  - Atrium Medisch Centrum Brunssum, Brunssum
  - Sint Antonius Ziekenhuis Nieuwegein, Nieuwegein
  - Refaja ziekenhuis, Stadskanaal
  - Medisch Centrum, Westeinde
- Norway (5):
  - Markeveien Spesialistpraksis, Bergen
  - Spesiallegetjenesten AS, Jessheim
  - Betanien Spesialistsenter, Oslo
  - Sykehuset Asker of Baerum HF, Rud
  - Forskningsstiftelsen Hjertelaget, Stravanger
- Poland (8):
  - Bydgoskie Centrum Diabetologii i Endokrynologii, Bydgoszcz
  - Oddzial Chorob Wewnetrznych, Częstochowa
  - NZOZ "Diab-Endo-Met", Krakow
  - Poradnia Diabetologiczna, Lodz
  - Poradnia Diabetologiczna, Lublin
  - Oddzial Chorob Wewnetrznych, Mielec
  - Oddzial Chorob Wewnetrznych i Diabetologii, Warsaw
  - Wojewodzka Poradnia dla Chorych na Cukrzyce, Warsaw
- Portugal (4):
  - Hospital Garcia de Orta-Servico de Endocrinologia, Almada
  - Centro Hospitalar de Coimbra, Coimbra
  - Associacao Protectora dos Diabeticos de Portugal, Lisbon
  - Hospital Geral de Santo Antonio, Porto
- Puerto Rico (6):
  - Universidad Central del Caribe, Bayamón
  - Hospital Alejandro Otero Lopez, Manatí
  - Dr. Luis Ruiz, Ponce
  - RCMI-Clinical Research Center, Rio Piedras
  - San Juan Health Center, San Juan
  - Centro de Endocrinologia del Este, Yabucoa
- Spain (5):
  - Hospital Vega Baja, Alicante
  - Hospital Doce de Octubre, Madrid
  - Hospital Gral de Mostoles, Madrid
  - Hospital Virgen de Valme, Seville
  - Hospital la Ribera, Alzira, Valencia
- Sweden (6):
  - Lundberglaboratoriet for diabetesforskning, Gothenburg
  - Medicinska kliniken, Helsingborg
  - Kliniska Forskningsenheren, Lund
  - Diabetesmottagningen, Intermedicinska kliniken, Stockholm
  - CME, M71, Stockholm
  - Enheten for metabol kontroll, Stockholm

REFERENCES:
- [Result] Heine RJ, Van Gaal LF, Johns D, Mihm MJ, Widel MH, Brodows RG; GWAA Study Group. Exenatide versus insulin glargine in patients with suboptimally controlled type 2 diabetes: a randomized trial. Ann Intern Med. 2005 Oct 18;143(8):559-69. doi: 10.7326/0003-4819-143-8-200510180-00006. PMID 16230722
- [Derived] Pencek R, Blickensderfer A, Li Y, Brunell SC, Anderson PW. Exenatide twice daily: analysis of effectiveness and safety data stratified by age, sex, race, duration of diabetes, and body mass index. Postgrad Med. 2012 Jul;124(4):21-32. doi: 10.3810/pgm.2012.07.2567. PMID 22913891
- [Derived] Fineman MS, Mace KF, Diamant M, Darsow T, Cirincione BB, Booker Porter TK, Kinninger LA, Trautmann ME. Clinical relevance of anti-exenatide antibodies: safety, efficacy and cross-reactivity with long-term treatment. Diabetes Obes Metab. 2012 Jun;14(6):546-54. doi: 10.1111/j.1463-1326.2012.01561.x. Epub 2012 Feb 10. PMID 22236356

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two patients were lost to follow-up after receiving study drug, and it is not known if they took at least one dose of the drug. For purposes of data analysis, these patients were classified as untreated.
Groups:
- Exenatide Arm: Exenatide subcutaneous injection twice daily for 26 weeks (5mcg for 4 weeks followed by 10mcg for 22 weeks)
- Insulin Glargine Arm: Insulin glargine subcutaneous injection once daily for 26 weeks (forced titration to target blood glucose level)
Period: Overall Study
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Started | 283 | 268
Received Treatment (Intent to Treat) | 282 | 267
Completed | 228 | 242
Not Completed | 55 | 26
Not completed — Adverse Event | 27 | 2
Not completed — Lost to Follow-up | 5 | 7
Not completed — Patient Decision | 8 | 4
Not completed — Physician Decision | 1 | 2
Not completed — Protocol Violation | 10 | 11
Not completed — Loss of Glucose Control | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide Arm | Insulin Glargine Arm | Total
Number analyzed (Participants) | 282 | 267 | 549
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.80 (8.82) | 57.96 (9.46) | 58.91 (9.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 116 | 243
  Male | 155 | 151 | 306

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Hemoglobin (HbA1c)
Description: Change in HbA1c from baseline to week 26
Time Frame: Baseline, week 26
Population: Last Observation Carried Forward; Intent to Treat, computed from the patients having both baseline and post baseline data
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Number analyzed (Participants) | 275 | 260
percentage
  Baseline HbA1c | 8.13 (0.07) | 8.19 (0.07)
  Change in HbA1c at week 26 | -1.00 (0.06) | -1.05 (0.06)
Statistical Analysis 1: Comparison: Exenatide Arm vs Insulin Glargine Arm; Test type: Non-Inferiority or Equivalence — Pre-specified non-inferiority margin was 0.4% (i.e., noninferiority is demonstrated if the upper limit of a two-sided 95% confidence interval for the difference in change in HbA1c between exenatide and insulin glargine is less than 0.4%.); p = 0.4602, ANCOVA; Mean Difference (Final Values) = 0.05, 95% CI [-0.09 to 0.20]

2. Secondary Outcome: Percentage of Patients Achieving HbA1c <=7%
Description: Percentage of patients in each arm who had HbA1c >7% at baseline and had HbA1c <=7% at week 26 (percentage = [number of subjects with HbA1c <=7% at week 26 divided by number of subjects with HbA1c >7% at baseline] * 100%).
Time Frame: 26 weeks
Population: Last Observation Carried Forward; Intent to Treat
Measure: Number; unit: percentage of participants
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Number analyzed (Participants) | 282 | 267
percentage of participants | 46.43 | 48.03
Statistical Analysis 1: Comparison: Exenatide Arm vs Insulin Glargine Arm; Test type: Superiority or Other; p = 0.7839, Fisher Exact

3. Secondary Outcome: Change in Body Weight
Description: Change in body weight from baseline to week 26
Time Frame: Baseline, week 26
Population: Intent to Treat
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Number analyzed (Participants) | 231 | 244
kg
  Baseline body weight | 88.42 (1.16) | 89.25 (1.20)
  Change in body weight at week 26 | -2.32 (0.21) | 1.75 (0.21)
Statistical Analysis 1: Comparison: Exenatide Arm vs Insulin Glargine Arm; Test type: Superiority or Other; p < 0.0001, ANCOVA

4. Secondary Outcome: Change in Fasting Serum Glucose
Description: Change in fasting serum glucose from baseline to week 26
Time Frame: Baseline, week 26
Population: Last Observation Carried Forward; Intent to Treat
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Number analyzed (Participants) | 258 | 245
mmol/L
  Baseline fasting serum glucose | 10.27 (0.21) | 10.46 (0.21)
  Change in fasting serum glucose at week 26 | -1.22 (0.19) | -2.86 (0.19)
Statistical Analysis 1: Comparison: Exenatide Arm vs Insulin Glargine Arm; Test type: Superiority or Other; p < 0.0001, ANCOVA

5. Secondary Outcome: Change in 7-point Self-monitored Blood Glucose (SMBG) Profile
Description: Change in 7-point (pre-breakfast, 2 hour post breakfast, pre-lunch, 2 hour post lunch, pre-dinner, 2 hour post dinner, 0300 hours) SMBG profile from baseline to week 26
Time Frame: Baseline, week 26
Population: Last Observation Carried Forward; Intent to Treat
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Number analyzed (Participants) | 282 | 267
mmol/L
  Pre-breakfast: Baseline SMBG | 9.47 (0.169) | 9.50 (0.173)
  Pre-breakfast: Change in SMBG at week 26 | -1.25 (0.130) | -2.56 (0.132)
  2hr post breatfast: Baseline SMBG | 12.51 (0.220) | 12.36 (0.226)
  2hr post breakfast: Change in SMBG at week 26 | -3.77 (0.171) | -2.86 (0.174)
  Pre-lunch: Baseline SMBG | 9.61 (0.218) | 9.47 (0.224)
  Pre-lunch: Change in SMBG at week 26 | -1.50 (0.156) | -1.93 (0.158)
  2hr post lunch: Baseline SMBG | 11.15 (0.222) | 10.96 (0.226)
  2hr post lunch: Change in SMBG at week 26 | -1.68 (0.173) | -1.69 (0.176)
  Pre-dinner: Baseline SMBG | 9.46 (0.211) | 9.35 (0.216)
  Pre-dinner: Change in SMBG at week 26 | -1.15 (0.156) | -1.72 (0.159)
  2hr post dinner: Baseline SMBG | 11.17 (0.206) | 11.49 (0.211)
  2hr post dinner: Change in SMBG at week 26 | -3.06 (0.172) | -1.65 (0.175)
  3:00 AM: Baseline SMBG | 9.02 (0.189) | 9.36 (0.192)
  3:00 AM: Change in SMBG at week 26 | -1.05 (0.169) | -1.97 (0.169)

6. Secondary Outcome: Percentage of Patients With Hypoglycemic Events
Description: Percentage of patients who experienced at least one episode of hypoglycemia at any point during the 26 week Parent Study (incidence of hypoglycemia = number of patients who experienced at least one episode of hypoglycemia at any point during the 26 week Parent Study divided by the total number of patients who participated in the 26 week Parent Study
Time Frame: 26 weeks
Population: Intent to Treat
Measure: Number; unit: percentage of participants
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Number analyzed (Participants) | 282 | 267
percentage of participants | 55.32 | 59.93
Statistical Analysis 1: Comparison: Exenatide Arm vs Insulin Glargine Arm; Test type: Superiority or Other; p = 0.3002, Fisher Exact

7. Secondary Outcome: Change in Rate of Hypoglycemic Events
Description: Change in rate of hypoglycemic events per 30 days per patient from baseline to week 26
Time Frame: Baseline, week 26
Population: Intent to Treat
Measure: Least Squares Mean (Standard Error); unit: events per 30 days per patient
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Number analyzed (Participants) | 282 | 267
events per 30 days per patient
  Baseline event rate | 0.09 (0.04) | 0.11 (0.04)
  Change in event rate at week 26 | 0.23 (0.06) | 0.29 (0.06)
Statistical Analysis 1: Comparison: Exenatide Arm vs Insulin Glargine Arm; Test type: Superiority or Other; p = 0.3385, ANCOVA

ADVERSE EVENTS:
Arm/Group | Exenatide Arm | Insulin Glargine Arm
Serious Adverse Events (participants affected / at risk) | 8 | 10
Other Adverse Events (participants affected / at risk) | 226 | 160
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Exenatide Arm | Insulin Glargine Arm
Hypertension (Vascular disorders) | 2/282 | 0/267
Alanine aminotransferase increased (Investigations) | 0/282 | 1/267
Angioneurotic edema (Skin and subcutaneous tissue disorders) | 0/282 | 1/267
Atrial fibrillation (Cardiac disorders) | 1/282 | 0/267
Calculus ureteric (Renal and urinary disorders) | 0/282 | 1/267
Cholelithiasis (Hepatobiliary disorders) | 1/282 | 0/267
Coronary artery atherosclerosis (Cardiac disorders) | 1/282 | 0/267
Coronary artery disease (Cardiac disorders) | 1/282 | 0/267
Dermatofibrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/282 | 0/267
Erysipelas (Infections and infestations) | 0/282 | 1/267
Humerus fracture (Injury, poisoning and procedural complications) | 0/282 | 1/267
Major depression (Psychiatric disorders) | 0/282 | 1/267
Metrorrhagia (Reproductive system and breast disorders) | 0/282 | 1/267
Non-cardiac chest pain (General disorders) | 0/282 | 1/267
Pancreatitis acute (Gastrointestinal disorders) | 0/282 | 1/267
Seroma (Injury, poisoning and procedural complications) | 1/282 | 0/267
Syncope (Nervous system disorders) | 0/282 | 1/267
Tachyarrhythmia (Cardiac disorders) | 1/282 | 0/267
Vomiting (Gastrointestinal disorders) | 1/282 | 0/267
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Exenatide Arm | Insulin Glargine Arm
Nausea (Gastrointestinal disorders) | 161/282 | 23/267
Vomiting (Gastrointestinal disorders) | 49/282 | 10/267
Headache (Nervous system disorders) | 25/282 | 23/267
Nasopharyngitis (Infections and infestations) | 22/282 | 24/267
Diarrhea (Gastrointestinal disorders) | 24/282 | 8/267
Upper respiratory tract infection (Infections and infestations) | 15/282 | 13/267
Back pain (Musculoskeletal and connective tissue disorders) | 17/282 | 8/267
Influenza (Infections and infestations) | 7/282 | 15/267
Dizziness (Nervous system disorders) | 15/282 | 6/267
Hypoglycemia (Metabolism and nutrition disorders) | 156/282 | 160/267

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days